CLINICAL TRIAL: NCT01206816
Title: An Open Label Phase I Dose Escalation Trial of Intravenous BI 6727 in Combination With Oral BIBW 2992 in Patients With Advanced Solid Tumours With Repeated Administration in Patients With Clinical Benefit
Brief Title: An Open Label Phase I Dose Escalation Trial of Intravenous BI 6727 (Volasertib)in Combination With Oral BIBW 2992 (Afatinib) in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 1230.20; 2010-019437-97 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BI 6727; Afatinib

ARMS (1):
- two experimental arms (Experimental): patients receive increasing doses of BI 6727 in combination with increasing doses of BIBW 2992
  Interventions: Drug: BI 6727 + BIBW 2992

INTERVENTIONS:
Drug: BI 6727 + BIBW 2992 — BI 6727 administered i.v. every 21 days + BIBW 2992 given orally once a day

SUMMARY:
The primary objective of the current study is to investigate the Maximum Tolerated Dose (MTD) in terms of safety and tolerability of the combination of BI 6727 with BIBW 2992, in patients with advanced or metastatic solid tumours. Dosages of both BI 6727 and BIBW 2992 will be varied to establish the MTD of the combination. Two combination treatment schedules will be tested, the MTD of each combination will be determined.

Secondary objectives are the exploration of pharmacokinetics, overall safety and preliminary efficacy.

ELIGIBILITY:
Inclusion criteria:

* Patients with histologically or cytologically confirmed diagnosis of advanced, non resectable and/or metastatic, relapsed or refractory solid tumours not amenable to standard therapy and for whom no therapy of proven efficacy exists
* Eastern Cooperative Oncology Group performance score 0 - 2
* Recovery from clinically significant toxicities from previous systemic anti-cancer therapies or radiotherapy

Exclusion criteria:

* Serious illness, concomitant non-oncological disease or mental problem considered by the investigator to be incompatible with participation to the trial
* Known hypersensitivity to the trial drugs or their excipients
* Treatment with any other investigational drug or active participation in any other interventional trial within 28 days before first administration of trial drug(s) or concomitantly with this trial
* Major surgery or radiotherapy within 28 days before start of therapy or concomitantly with this trial
* Systemic anti-cancer therapy within 28 days before start of therapy or concomitantly with this trial
* Requirements for treatment with any of the prohibited concomitant medications
* Active infectious disease or known HIV I/II infection
* Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhoea
* Active brain metastases
* History or presence of cardiovascular abnormalities deemed clinically relevant by the investigator
* Cardial left ventricular function with resting ejection fraction < 50%
* Inadequate hepatic, renal and haematologic organ function
* QT prolongation deemed clinically relevant by the investigator
* Active alcohol or drug abuse
* Women of childbearing potential and men who are able to father a child unwilling to use a medically acceptable method of contraception during the trial and 28 days thereafter
* Pregnancy or breast-feeding
* Patients unable to comply with the protocol
* Patients with known pre-existing interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-10-04 (Actual); Primary Completion 2012-11-15 (Actual); Study Completion 2012-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Belgium (3):
  - 1230.20.32001 Boehringer Ingelheim Investigational Site, Brussels
  - 1230.20.32003 Boehringer Ingelheim Investigational Site, Edegem
  - 1230.20.32002 Boehringer Ingelheim Investigational Site, Ghent

REFERENCES:
- [Derived] Machiels JP, Peeters M, Herremans C, Surmont V, Specenier P, De Smet M, Pilz K, Strelkowa N, Liu D, Rottey S. A phase I study of volasertib combined with afatinib, in advanced solid tumors. Cancer Chemother Pharmacol. 2015 Oct;76(4):843-51. doi: 10.1007/s00280-015-2860-2. Epub 2015 Sep 8. PMID 26349473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Aspartate amino transferase (AST) ; Alanine amino transferase (ALT) and Eastern Cooperative Oncology Group (ECOG).
Pre-assignment Details: This is a Phase 1, open label, non randomised and dose escalation trial. There was no control group. The Combination of Volasertib and Afatinib to be investigated in two treatment schedules (A & B). In Schedule B the starting doses will be depend on the outcome of the MTD determination from treatment schedule A.
Groups:
- Volasertib150 mg+Afatinib 30 mg (Schedule A): Schedule A : Volasertib (Vol) 150 mg on Day 1 and afatinib (aftb) 30 mg from Day 2 to Day 21.
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
- Volasertib 225 mg+Afatinib 30 mg (Schedule A): Schedule A : Volasertib 225 mg on Day 1 and afatinib 30 mg from Day 2 to Day 21.
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
- Volasertib 300 mg+Afatinib 30 mg (Schedule A): Schedule A :Volasertib 300 mg on Day 1 and afatinib 30 mg from Day 2 to Day 21.
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
- Volasertib 300 mg+Afatinib 40 mg (Schedule A): Schedule A :Volasertib 300 mg on Day 1 and afatinib 40 mg from Day 2 to Day 21.
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
- Volasertib 300 mg+Afatinib 50 mg (Schedule B): Schedule B: Volasertib 300 mg on Day 1 and afatinib 50 mg pulsed from Day 2 to Day 6 (no administration of afatinib from Day 7 to 21).
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
- Volasertib 300 mg+Afatinib 70 mg (Schedule B): Schedule B: Volasertib 300 mg on Day 1 and afatinib 70 mg pulsed from Day 2 to Day 6 (no administration of afatinib from Day 7 to 21).
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
- Volasertib 300 mg+Afatinib 90 mg (Schedule B): Schedule B : Volasertib 300 mg on Day 1 and afatinib 90 mg pulsed from Day 2 to Day 6 (no administration of afatinib from Day 7 to 21).
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
Period: Overall Study
Arm/Group | Volasertib150 mg+Afatinib 30 mg (Schedule A) | Volasertib 225 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 40 mg (Schedule A) | Volasertib 300 mg+Afatinib 50 mg (Schedule B) | Volasertib 300 mg+Afatinib 70 mg (Schedule B) | Volasertib 300 mg+Afatinib 90 mg (Schedule B)
Started | 3 (Started=Treated) | 3 (Started=Treated) | 20 (Started=Treated) | 3 (Started=Treated) | 3 (Started=Treated) | 19 (Started=Treated) | 6 (Started=Treated)
Completed | 0 | 0 | 0 (1pt dist.due to 'Other AE' for vol& since 'other' from aftb.1pt 'PD' for vol& since,'DLT' from aftb) | 0 (1pt discontinue (dist.)due to 'PD' for vol.& since, 'Other AE' from aftb) | 0 | 0 (1pt dist. due to 'PD' for vol & since, 'Other AE' from aftb) | 0 (1pt dist. due to 'other AE' & 1pt 'other' for vol & since,'PD' from aftb.)
Not Completed | 3 | 3 | 20 | 3 | 3 | 19 | 6
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 3 | 3 | 13 | 3 | 3 | 16 | 3
Not completed — Other AE | 0 | 0 | 4 | 0 | 0 | 3 | 2
Not completed — other than stated above | 0 | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All 57 patients who received at least 1 dose of volasertib and afatinib were included in the treated set
Groups:
- Volasertib 300 mg+Afatinib 30 mg (Schedule A): Schedule A : Volasertib 300 mg on Day 1 and afatinib 30 mg from Day 2 to Day 21.
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
- Volasertib 300 mg+Afatinib 40 mg (Schedule A): Schedule A : Volasertib 300 mg on Day 1 and afatinib 40 mg from Day 2 to Day 21.
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
- Total: Total of all reporting groups
Arm/Group | Volasertib150 mg+Afatinib 30 mg (Schedule A) | Volasertib 225 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 40 mg (Schedule A) | Volasertib 300 mg+Afatinib 50 mg (Schedule B) | Volasertib 300 mg+Afatinib 70 mg (Schedule B) | Volasertib 300 mg+Afatinib 90 mg (Schedule B) | Total
Number analyzed (Participants) | 3 | 3 | 20 | 3 | 3 | 19 | 6 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (18.7) | 48.7 (6.1) | 54.5 (7.6) | 57.0 (10.8) | 62.3 (4.9) | 61.9 (9.3) | 64.2 (6.0) | 58.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 10 | 2 | 0 | 10 | 3 | 28
  Male | 1 | 2 | 10 | 1 | 3 | 9 | 3 | 29
ECOG at screening [Count of Participants; unit: Participants] — the Eastern Cooperative Oncology Group (ECOG) performance score was between 0 and 2. 0: Normal activity. Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2=Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours;
  Participants
    0 | 1 | 2 | 8 | 1 | 1 | 5 | 2 | 20
    1 | 2 | 1 | 11 | 2 | 2 | 13 | 3 | 34
    2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
Tumour classification [Count of Participants; unit: Participants]
  Head & neck cancers | 0 | 1 | 6 | 1 | 0 | 0 | 1 | 9
  Non small cell lung | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Gastrointest. tract | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Colorectal (col/rec) | 1 | 0 | 6 | 0 | 2 | 12 | 2 | 23
  Anal region | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Pancreas | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 5
  Biliary tree | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Genitourinary system | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Ureter | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Gynecologic cancers | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Cancers of breast | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 5
  Soft tissue/oss sarc | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Other | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 4
  Missing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: MTD was defined on the basis of DLTs occuring during Cycle 1 of the dose escalation part in each of the 2 treatment schedules. DLTs were defined as drug related based on Common Terminology Criteria for AE's (CTCAE) Grade(G) :1) G4 neutropenia (ANC, including bands, <500/mm³) for more than 7 days, 2) G3 or 4 neutropenia associated with fever >38.5° C (febrile neutropenia),3) Neutropenic infection G ≥3, 4) G4 thrombocytopenia or G3 thrombocytopenia associated with bleeding requiring whole blood transfusion.5) Non-haematological G ≥3 toxicity excluding: (a) untreated G3 diarrhoea, (b) untreated G3 nausea and/or vomiting, (c) untreated G3 rash. 6) G2 increase in AST and/or ALT in conjunction with an elevated bilirubin level of G ≥2, 7) G2 nausea and/or vomiting despite optimal supportive/antiemetic treatment for at least 7consecutive days. 8) G2 diarrhoea for 2 or more consecutive days despite antidiarrhoeal medication/hydration, 9) Decrease in left ventricular function G ≥2.
Time Frame: 22 Days
Population: Treated Set (TS)
Measure: Number; unit: participants
Arm/Group | Volasertib150 mg+Afatinib 30 mg (Schedule A) | Volasertib 225 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 40 mg (Schedule A) | Volasertib 300 mg+Afatinib 50 mg (Schedule B) | Volasertib 300 mg+Afatinib 70 mg (Schedule B) | Volasertib 300 mg+Afatinib 90 mg (Schedule B)
Number analyzed (Participants) | 3 | 3 | 20 | 3 | 3 | 19 | 6
participants | 0 | 0 | 3 | 2 | 0 | 5 | 2

2. Primary Outcome: Maximum Tolerable Dose (MTD) of Two Combination Therapy of Volasertib and Afatinib.
Description: Maximum Tolerable Dose (MTD) was determined by dose escalation for volasertib and afatinib. The "3 + 3 design with de-escalation" for both the Schedules A and B. Patients were sequentially allocated to the dose cohorts. Apart from allocation to the treatment schedules, escalation and/or de-escalation to determine the MTD occurred independently within the 2 dose schedules. Cohorts of 3 patients were to be treated at the starting dose levels according to the treatment schedule. Before entering patients at a higher dose level, all patients at the previous dose level combination had to complete at least the initial cycle of 21 days.
Time Frame: MTD was assessed during the first cycle of combination of Volasertib and Afatinib therapy (22 days)
Population: Treated Set (TS)
Measure: Number; unit: mg
Groups:
- Volasertib in Combination With Afatinib (Schedule A): The combination of Volasertib and Afatinib were investigated in two treatment schedules (A & B). In schedule A, Dose level 1: Volasertib 150 mg and afatinib 30 mg . Dose level 2: Volasertib 225 mg and afatinib 30 mg. Dose level 3: Volasertib 300 mg and afatinib 30 mg. Dose level 4: Volasertib 300 mg and afatinib 40 mg. In schedule B , Dose level 1: Volasertib 300 mg and afatinib 50 mg. Dose level 2: Volasertib 300 mg and afatinib 70 mg. Dose level 3: Volasertib 300 mg and afatinib 90mg.
  In schedule A, Volasertib was infused on Day 1 and afatinib from Day 2 to Day 21. In schedule B, Volasertib on Day 1 and afatinib pulsed from Day 2 to Day 6 (no administration of afatinib from Day 7 to 21). Schedule B was depending on the outcome of the MTD determination from treatment schedule A.
- Volasertib in Combination With Afatinib (Schedule B): The combination of Volasertib and Afatinib were investigated in two treatment schedules (A & B). In schedule B , Dose level 1: Volasertib 300 mg and afatinib 50 mg. Dose level 2: Volasertib 300 mg and afatinib 70 mg. Dose level 3: Volasertib 300 mg and afatinib 90mg.
Arm/Group | Volasertib in Combination With Afatinib (Schedule A) | Volasertib in Combination With Afatinib (Schedule B)
Number analyzed (Participants) | 29 | 28
mg
  Volasertib | 300 | 300
  Afatinib | 30 | 70

3. Secondary Outcome: Number of Patients With Drug-related Adverse Events According to Common Terminology Criteria for Adverse Events (CTCAE) Criteria v 3.0
Description: Number of patients with investigator defined drug-related adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) criteria v 3.0
Time Frame: After the first drug administration until 28 days after the last drug administration, up to 413 days.
Population: Treated Set (TS)
Measure: Number; unit: participants
Arm/Group | Volasertib150 mg+Afatinib 30 mg (Schedule A) | Volasertib 225 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 40 mg (Schedule A) | Volasertib 300 mg+Afatinib 50 mg (Schedule B) | Volasertib 300 mg+Afatinib 70 mg (Schedule B) | Volasertib 300 mg+Afatinib 90 mg (Schedule B)
Number analyzed (Participants) | 3 | 3 | 20 | 3 | 3 | 19 | 6
participants | 3 | 3 | 18 | 3 | 3 | 19 | 6

4. Secondary Outcome: Number of Patients With Objective Response (OR)
Description: Objective tumor response based on response evaluation criteria in solid tumors (RECIST) version 1.1. OR is defined as complete response (CR) or partial response (PR).
  As Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by using appropriate radiology techniques: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Tumor assessment was performed at screening and at the end of every 3 treatment cycle (ie every 9 weeks of treatment).
Population: Treated Set (TS)
Measure: Number; unit: participants
Arm/Group | Volasertib150 mg+Afatinib 30 mg (Schedule A) | Volasertib 225 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 40 mg (Schedule A) | Volasertib 300 mg+Afatinib 50 mg (Schedule B) | Volasertib 300 mg+Afatinib 70 mg (Schedule B) | Volasertib 300 mg+Afatinib 90 mg (Schedule B)
Number analyzed (Participants) | 3 | 3 | 20 | 3 | 3 | 19 | 6
participants
  Yes | 1 | 0 | 1 | 0 | 0 | 0 | 0
  No | 2 | 3 | 17 | 3 | 3 | 15 | 6
  Unknown | 0 | 0 | 2 | 0 | 0 | 4 | 0

5. Secondary Outcome: Number of Patients With Best Overall Response.
Description: Best overall response based on response evaluation criteria in solid tumors (RECIST) version 1.1. Best overall response is defined as complete response, partial response, stable disease, progressive disease or not evaluable.
  As Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by using appropriate radiology techniques: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: Tumor assessment was performed at screening and at the end of every 3 treatment cycle (ie every 9 weeks of treatment).
Population: Treated Set (TS)
Measure: Number; unit: participants
Groups:
- Volasertib 300 mg+Afatinib 40 mg (Schedule A): Schedule A (Cycle 1):Volasertib 300 mg on Day 1 and afatinib 40 mg from Day 2 to Day 21.
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
Arm/Group | Volasertib150 mg+Afatinib 30 mg (Schedule A) | Volasertib 225 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 40 mg (Schedule A) | Volasertib 300 mg+Afatinib 50 mg (Schedule B) | Volasertib 300 mg+Afatinib 70 mg (Schedule B) | Volasertib 300 mg+Afatinib 90 mg (Schedule B)
Number analyzed (Participants) | 3 | 3 | 20 | 3 | 3 | 19 | 6
participants
  Complete response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Stable disease | 0 | 0 | 8 | 0 | 1 | 5 | 2
  Progressive disease | 2 | 3 | 8 | 3 | 2 | 10 | 4
  Not evaluable | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 2 | 0 | 0 | 4 | 0

6. Secondary Outcome: Number of Patients With Disease Control
Description: Disease control based on response evaluation criteria in solid tumors (RECIST) version 1.1. Patients who had a best overall tumour response of complete response (CR), partial response (PR) or stable disease (SD) were assessed to show disease control.
  As Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by using appropriate radiology techniques: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: Tumor assessment was performed at screening and at the end of every 3 treatment cycle (ie every 9 weeks of treatment).
Population: Treated Set (TS)
Measure: Number; unit: participants
Arm/Group | Volasertib150 mg+Afatinib 30 mg (Schedule A) | Volasertib 225 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 40 mg (Schedule A) | Volasertib 300 mg+Afatinib 50 mg (Schedule B) | Volasertib 300 mg+Afatinib 70 mg (Schedule B) | Volasertib 300 mg+Afatinib 90 mg (Schedule B)
Number analyzed (Participants) | 3 | 3 | 20 | 3 | 3 | 19 | 6
participants
  YES | 1 | 0 | 9 | 0 | 1 | 5 | 2
  NO | 2 | 3 | 9 | 3 | 2 | 10 | 4
  Unknown | 0 | 0 | 2 | 0 | 0 | 4 | 0

ADVERSE EVENTS:
Time Frame: After the first drug administration until 28 days after the last drug administration, upto 413 days.
Groups:
- Volasertib 300 mg+Afatinib 50 mg (Schedule B): Schedule B : Volasertib 300 mg on Day 1 and afatinib 50 mg pulsed from Day 2 to Day 6 (no administration of afatinib from Day 7 to 21).
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
- Volasertib 300 mg+Afatinib 70 mg (Schedule B): Schedule B : Volasertib 300 mg on Day 1 and afatinib 70 mg pulsed from Day 2 to Day 6 (no administration of afatinib from Day 7 to 21).
  Cycle 1 was completed after 21 days on Day 22. All subsequent cycles lasted 21 days. Patients that started a second cycle were to be co-administered with volasertib and afatinib on Day 1 of the second cycle. Afatinib was to be taken before the start of the volasertib infusion.
Arm/Group | Volasertib150 mg+Afatinib 30 mg (Schedule A) | Volasertib 225 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 30 mg (Schedule A) | Volasertib 300 mg+Afatinib 40 mg (Schedule A) | Volasertib 300 mg+Afatinib 50 mg (Schedule B) | Volasertib 300 mg+Afatinib 70 mg (Schedule B) | Volasertib 300 mg+Afatinib 90 mg (Schedule B)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 11/20 | 2/3 | 1/3 | 12/19 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 18/20 | 3/3 | 3/3 | 19/19 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib150 mg+Afatinib 30 mg (Schedule A) (N=3) | Volasertib 225 mg+Afatinib 30 mg (Schedule A) (N=3) | Volasertib 300 mg+Afatinib 30 mg (Schedule A) (N=20) | Volasertib 300 mg+Afatinib 40 mg (Schedule A) (N=3) | Volasertib 300 mg+Afatinib 50 mg (Schedule B) (N=3) | Volasertib 300 mg+Afatinib 70 mg (Schedule B) (N=19) | Volasertib 300 mg+Afatinib 90 mg (Schedule B) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Puncture site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib150 mg+Afatinib 30 mg (Schedule A) (N=3) | Volasertib 225 mg+Afatinib 30 mg (Schedule A) (N=3) | Volasertib 300 mg+Afatinib 30 mg (Schedule A) (N=20) | Volasertib 300 mg+Afatinib 40 mg (Schedule A) (N=3) | Volasertib 300 mg+Afatinib 50 mg (Schedule B) (N=3) | Volasertib 300 mg+Afatinib 70 mg (Schedule B) (N=19) | Volasertib 300 mg+Afatinib 90 mg (Schedule B) (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 7 | 1 | 1 | 9 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 8 | 2 | 0 | 8 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 7 | 1 | 0 | 9 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelids pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 7 | 0 | 0 | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 3 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 4 | 0 | 0 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 15 | 1 | 3 | 18 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 10 | 1 | 1 | 9 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Perianal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 8 | 1 | 0 | 8 | 4
Vomiting (Gastrointestinal disorders) | 2 | 0 | 7 | 1 | 2 | 5 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 2 | 3 | 11 | 2 | 1 | 14 | 3
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 4 | 1 | 0 | 3 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 4 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 3 | 1 | 1 | 5 | 1
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 3 | 2
Neutropenic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 3 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 11 | 2 | 1 | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 1 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 2 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 0 | 3 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 4 | 0 | 0 | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 0 | 0 | 4 | 2
Bladder irritation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 0 | 1 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 5 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 0 | 0 | 5 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0 | 1 | 4 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 5 | 0 | 1 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 4 | 0 | 0 | 1 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 8 | 2 | 1 | 7 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 1 | 0 | 1 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vasoconstriction (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.